CLINICAL TRIAL: NCT06513910
Title: Evaluating the Impact of Community-Based Mindfulness and Musical Programs on Psychiatric Measures, Social Music Study 2b.
Brief Title: Evaluating the Impact of Social Music
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000028866_b; 2R25MH071584-11 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Mental Health Issue; COVID-19
Keywords: Mindfulness; Meditation; Music
MeSH Terms: conditions — COVID-19 | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be screened, consented, and enrolled in dyads.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Component 2b. Social Music Study (Experimental): Investigators will assess the neural mechanisms of feelings of subjective connectedness during communal music listening and creating between dyads of subjects who are both familiar and unfamiliar with each other
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — Participants in dyads will be positioned across from each other while listening to various types of music (i.e. music that is harmonically-intact and music in which the harmonic content has been randomly scrambled).

SUMMARY:
Mental health vulnerability due to stress is increased in People of African Descent (PADs) in America due to disproportionate effects of racism, poverty, education, and criminal justice sentencing. Various meditation and mindfulness approaches have provided evidence of measured reductions in multiple negative dimensions of stress. However, the majority of these studies do not have an adequate representation of PADs or other marginalized groups and are not designed to be culturally relevant or community based. Music has been shown to alleviate multiple symptoms of stress and has been shown to be a preferred and effective support for meditation and mindfulness. However, its role in stress management in PADs engaged in meditation or mindfulness is seldom studied. This study aims to evaluate the effects of a virtual, community-based music mindfulness program on stress management in PAD community members with anxiety and depression during COVID19.

2b. Social Music Study: Investigators will assess the neural mechanisms of feelings of subjective connectedness during communal music listening and creating between dyads of subjects who are both familiar and unfamiliar with each other.

DETAILED DESCRIPTION:
The investigators also propose a study to investigate the effects of communal drumming in reducing anxiety and increasing connectedness within drum circle community. Investigators hypothesize that these intervention will lead to reductions in scores on stress scales and will provide preliminary data for studies evaluating these types of community programs as an adjunct to the standard of care.

Participants will be screened, consented, and enrolled in dyads in a paradigm in which they will be positioned across from each other while listening to various types of music (i.e. music that is harmonically-intact and music in which the harmonic content has been randomly scrambled).

Survey data will also be collected to assess variables such as musical experience, partner familiarity, perceived stress, etc.

ELIGIBILITY:
Inclusion Criteria:

* ages 16 and older

Exclusion Criteria:

* contraindications to functional Near Infrared Spectroscopy or Electroencephalography
* ages 15 and younger

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
EEG gamma and theta activity during music vs no music conditions | baseline measurements on day of study, during music vs no music conditions, and 30 minutes after music listening
  EEG gamma and theta activity measured by the Post Spectral Density measures in the gamma range (>30Hz) and theta (4-8Hz) frequency ranges during music vs no music conditions.

SECONDARY OUTCOMES:
Mean score subjective rating of social connection during session | baseline measurements on day of study, during music vs no music conditions, and 30 minutes after music listening
  Rating of subjective connectedness will be assessed using a Likert scale with total score range from 1-5, with higher scores indicating more connectedness.

CONTACTS AND LOCATIONS:
Overall Officials: AZA Allsop, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - BLOOM, New Haven, Connecticut
  - Musical Intervention Studios, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified, aggregate data will be shared through pre-prints, publications, and community town hall meetings.